CLINICAL TRIAL: NCT02671227
Title: Effects of Addition of Magnesium Sulfate in Spinal Anesthesia on Surgeon Satisfaction and Postoperative Pain in Gynecologic Laparoscopic Surgeries.
Brief Title: Intrathecal Mg in Gynecologic Laparoscopic Surgeries.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, khaled salah mohamed, lecturer of anaesthesia and ICU, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: intrathecal Mg in gyne. lap.
Record Dates: First submitted 2016-01-24; First posted 2016-02-02 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-08

CONDITIONS: Gynecologic Laparoscopic Surgery

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intrathecal bupivacaine + Mg sulfate (Active Comparator): intrathecal bupivacaine 15 mg + intrathecal Mg sulfate 50 mg. in gynecologic laparoscopic surgeries.
  Interventions: Drug: intrathecal Mg sulfate.; Drug: intrathecal bupivacaine 15 mg.
- intrathecal bupivacaine (Active Comparator): intrathecal bupivacaine 15 mg in gynecologic laparoscopic surgeries.
  Interventions: Drug: intrathecal bupivacaine 15 mg.

INTERVENTIONS:
Drug: intrathecal Mg sulfate. — intrathecal Mg sulfate 50 mg.
  Arms: intrathecal bupivacaine + Mg sulfate
Drug: intrathecal bupivacaine 15 mg. — intrathecal bupivacaine 15 mg.

SUMMARY:
The investigators aim to investigate the differences between intrathecal Bupivacaine + Mg sulfate in spinal anesthesia versus Bupivacaine on surgeon satisfaction and postoperative pain in gynecologic laparoscopic surgeries.

DETAILED DESCRIPTION:
The investigators aim to investigate the differences between intrathecal Bupivacaine + Mg sulfate in spinal anesthesia versus Bupivacaine on surgeon satisfaction, patient satisfaction and postoperative pain in gynecologic laparoscopic surgeries.

ELIGIBILITY:
Inclusion Criteria:

* female patient.
* more than 18 years.
* undergoing elective gynecologic laparoscopic surgeries.

Exclusion Criteria:

* allergy to local anesthesia.
* contraindication to spinal anesthesia.
* Significant cardiac, liver or renal dysfunction.
* Inability to informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
surgeon satisfaction (scale from 1 to 10) . | intraoperative (from beginning of the gynecologic laparoscopic procedure till the end of the procedure).
  surgeon satisfaction (scale from 1 to 10) as 1 is worst and 10 is best.

SECONDARY OUTCOMES:
postoperative pain management (VAS score). | postoperative for 6 hours.
  Visual Analog Scale (VAS score).

CONTACTS AND LOCATIONS:
Locations (1):
- Asiut university hospital, Asiut, Egypt

IPD SHARING:
Plan to Share IPD: Yes